CLINICAL TRIAL: NCT05122507
Title: Liquid Biopsy of Head and Neck Cancer Patients in Blood and Saliva
Acronym: KOHACIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: KOHACIN
Record Dates: First submitted 2021-10-25; First posted 2021-11-16 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Liquid Biopsy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue, EDTA blood plasma, serum, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective study for therapy monitoring of locally advanced and metastatic head and neck cancer patients by detection of circulating tumor nucleic acids in peripheral blood and saliva

DETAILED DESCRIPTION:
Clinical examination including imaging and - if necessary - tissue biopsy sampling - is the current clinical standard in therapy monitoring of metastatic head and neck tumors. This includes both the initial diagnosis, the assessment of the therapeutic response during ongoing chemotherapy / radiochemotherapy and follow-up care with the aim of detecting recurrences at an early stage. The detection of circulating nucleic acids as well as proteins in the peripheral blood and saliva could represent a minimally invasive and exact method for the assessment of the tumor burden, for the early detection of recurrences and for the individual assessment of the therapy response in patients with head and neck cancer. The present study aims to evaluate the value of tumor-specific nucleic acids and proteins in peripheral blood and saliva as possible biomarkers for minimally invasive therapy monitoring of head and neck tumors. For this purpose, Next Generation Sequencing (NGS), ELISA and quantitative polymerase chain reaction (PCR) methods are used as diagnostic methods. NGS initially enables the creation of a genetic profile of the primary tumor with targeted massive parallel sequencing of frequently mutated genes in head and neck tumors. The amount of nucleic acids in the peripheral blood and saliva is then quantified by means of digital PCR with the aid of specifically designed digital PCR assays. In addition, tumor-associated nucleic acids and proteins in the primary tumor, blood and saliva are examined. The aim is to examine if the amount of tumor specific circulating nucleic acids and the concentration of protein biomarkers found in the blood and saliva are associated with the response to treatment, early detection of recurrence, and the overall prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck squamous cell carcinoma (HNSCC)
* Written informed consent

Exclusion Criteria:

* Neoplasms other than HNSCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for HNSCC at Klinikum rechts der Isar der Technischen Universität München
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Early recurrence detection lead time | Assessed up to 24 months
  Lead time is defined as time between liquid-biopsy based recurrence detection and clinical recurrence or progression.

SECONDARY OUTCOMES:
Recurrence-free survival | Assessed up to 24 months
  Recurrence-free survival
Overall survival | Assessed up to 24 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Irina Kerle, MD, Principal Investigator — Technical University of Munich; Markus Wirth, MD, Principal Investigator — Technical University of Munich; Christof Winter, MD, PhD, Principal Investigator — Technical University of Munich
Locations (1):
- Klinikum rechts der Isar der Technischen Universität München, Munich, Germany

IPD SHARING:
Plan to Share IPD: No